CLINICAL TRIAL: NCT05017220
Title: The Effects of Nature-based Sensory Stimulation on Pain in Women With Fibromyalgia: A Randomised Controlled Trial
Brief Title: Nature-based Sensory Stimulation on Pain Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Principal Investigator / Associate professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NBS in chronic pain patients
Record Dates: First submitted 2021-07-05; First posted 2021-08-23 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Nature-based activities; Pain dimensions; Multisensory stimulation; Quantitative sensory testing
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-based stimulation program (Experimental): Participants will receive a single intervention with a duration of 30 minutes based on a multisensorial nature-based stimulation
  Interventions: Other: Nature-based sensory stimuli
- Control intervention (Other): Participants will be involved in a placebo task for 30 minutes
  Interventions: Other: Control group intervention

INTERVENTIONS:
Other: Nature-based sensory stimuli — A program based on stimulation using nature-based sensory stimuli will be implemented
  Other Names: Biogenic sensory stimuli
  Arms: Nature-based stimulation program
Other: Control group intervention — An activity based on a placebo intervention will be implemented
  Arms: Control intervention

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a single session intervention based on a nature-based stimulation program in patients with fibromyalgia

DETAILED DESCRIPTION:
All participants will continue to receive their usual pharmacological treatment as previously established by the Andalusian Public Health System. The intervention will comprise interaction tasks with biotic and abiotic agents for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia syndrome (ACR criteria 2016).
* Chronic widespread musculoskeletal pain symptoms (>1 location using the Widespread Pain Index).
* High-intensity pain (VAS ≥ 4), at least 3 days a week for the previous 3 months.
* If currently taking analgesic or psychotropic medications, they had to be stabilised for four or more weeks before the study enrolment
* Over 18 and less than 65 years old (labour active).
* Ability to speak and understand English or Spanish.

Exclusion Criteria:

* Acute or temporal pain
* Severe cognitive impairment, detected by the Mini-Mental State Examination (score <24 out of 30 points)
* Severe mental disorders in acute phase or symptomatic phase
* Behavioural alterations as this may interfere in their participation
* Severe intellectual disability
* Other severe or medically unstable diseases interfering with the project participation
* Co-occurrence of neuropathic pain
* Other disorders that may cause pain
* Pregnant or breast-feeding
* Drug abuse within the past year.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline pain intensity after 30 minutes
  Clinical pain intensity assessed by an 11-points Numeric Rating Scale (NRS-11) ranging from 0 to 10
Cold pain thresholds | Change from baseline cold pain thresholds after 30 minutes
  Cold pressor test will be used
Punctate mechanical hyperalgesia | Change from baseline mechanical hyperalgesia after 30 minutes
  Semmes-Weinstein monofilament (Aesthesio® Precise Tactile Sensory Evaluator, DanMic Global, LLC, San Jose, CA, USA) calibrated to bend at 300 gm (2940 mN; size 6.65; 0.1143 cm in diameter) of pressure with a response-dependent method will be used
Wind-up phenomenon | Change from baseline temporal summation of pain perception after 30 minutes
  Wind-up is a frequency- and intensity-dependent increase in the excitability of dorsal horn neuron that results in a temporal summation of pain perception.
Pressure pain thresholds | Change from baseline pressure pain thresholds after 30 minutes
  The minimum pressure force which induces pain when pressure is applied on tissues is regarded as the pressure pain threshold

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Health Sciences, Granada
  - Universidad de Granada, Granada

IPD SHARING:
Plan to Share IPD: No